CLINICAL TRIAL: NCT04178902
Title: A First In Human Study of the MCL-1 Inhibitor, ABBV-467
Brief Title: A Study of the Safety and Tolerability of ABBV-467 in Adult Participants With Relapsed/Refractory (R/R) Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M19-025; 2018-003744-24 (EudraCT Number)
Record Dates: First submitted 2019-11-25; First posted 2019-11-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Multiple Myeloma (MM); Cancer
Keywords: Multiple Myeloma (MM); Relapse/Refractory; Cancer; ABBV-467
MeSH Terms: conditions — Multiple Myeloma; Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part A: ABBV-467 Dose Escalation (Experimental): ABBV-467 administered by intravenous (IV) infusion at various doses until a recommended phase 2 dose is determined.
  Interventions: Drug: ABBV-467
- Part B: ABBV-467 Dose Expansion (Experimental): ABBV-467 administered by intravenous (IV) infusion at recommended phase 2 dose as identified in Part A.
  Interventions: Drug: ABBV-467

INTERVENTIONS:
Drug: ABBV-467 — Intravenous (IV) Infusion

SUMMARY:
This first-in-human study will evaluate the safety and tolerability of ABBV-467 in adult participants with relapsed/refractory multiple myeloma (MM).

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of multiple myeloma (MM).
* Measurable disease defined as at least 1 of the following:

  * Serum monoclonal protein >= 1g/dL.
  * Urine M-protein >= 200mg/24 hours.
  * Serum immunoglobulin free light chain (FLC) >= 10 mg/dL (100 mg/L), provided serum FLC ratio is abnormal.
* Relapsed after or are refractory or intolerant to all established MM therapies that are both known to provide clinical benefit and locally available.
* Received at least 3 prior lines of therapy including 1 or more immunomodulatory agents, 1 or more proteasome inhibitors, and 1 or more anti-CD38 monoclonal antibodies.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Adequate hematologic, renal and hepatic function as described in the protocol.
* Echocardiogram with ejection fraction >= 50% and no other clinically significant findings that would increase the participant's susceptibility to cardiac toxicity.

Exclusion Criteria:

* Prior exposure to any targeted myeloid cell leukemia-1 (MCL-1) inhibitor.
* Antineoplastic therapy (including any cytotoxic, targeted and/or investigational therapy; but not including corticosteroids), within 28 days or 5 half-lives, whichever is shorter, prior to the first dose of study drug and through the last dose of study drug.
* Autologous stem cell transplant within 90 days prior to start of study drug.
* Allogenic stem cell transplant within 180 days prior to start of study drug.
* History of acute or chronic pancreatitis.
* Significant unresolved liver disease.
* History of hepatitis B or human immunodeficiency virus (HIV) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Up to approximately 24 months after first dose of study drug
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator will assess the relationship of each event to the use of study drug as being of reasonable possibility or no reasonable possibility. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent events (TEAEs/TESAEs) are defined as any event that began or worsened in severity after the first dose of study drug.
Change in Vital Signs | Baseline (Week 0) through approximately 24 months after first dose of study drug
  Change in vital signs like systolic and diastolic blood pressure will be assessed.
Change in Electrocardiogram (ECG) | Baseline (Week 0) through approximately 24 months after first dose of study drug
  12-lead resting ECGs will be recorded. Parameters include RR interval, PR interval, QT interval, and QRS duration.
Change in Cardiac Enzyme Levels | Baseline (Week 0) through approximately 24 months after first dose of study drug
  Change in cardiac enzyme levels will be recorded.
Incidence of Abnormal Clinical Laboratory Test Results | Baseline (Week 0) through approximately 24 months after first dose of study drug
  Number of participants with incidence of abnormal clinical laboratory test results like hematology will be assessed.
Maximum Observed Plasma Concentration (Cmax) | Up to approximately Day 197
  Maximum Plasma Concentration (Cmax) of ABBV-467.
Terminal Phase Elimination Half-life (t1/2) | Up to approximately Day 197
  Terminal phase elimination half-life (t1/2) of ABBV-467
Area Under the Plasma Concentration-Time Curve (AUCt) | Up to approximately Day 197
  AUC from time 0 to time of last measurable concentration of ABBV-467.
Area Under the Plasma Concentration-Time Curve (AUC0-infinity) | Up to approximately Day 197
  AUC from time 0 to infinity of ABBV-467.
Clearance of ABBV-467 | Up to approximately Day 197
  Clearance of ABBV-467.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 24 months after first dose of study drug
  ORR evaluated per adapted International Myeloma Working Group (IMWG) criteria and defined as partial response (PR) + very good partial response (VGPR) + complete remission (CR) + stringent complete response (sCR).
Clinical Benefit Rate (CBR) | Up to approximately 24 months after first dose of study drug
  CBR evaluated per adapted International Myeloma Working Group (IMWG) criteria and is defined as minimal response (MR) + PR + VGPR + CR + sCR.
Duration of Response (DOR) | Up to approximately 24 months after first dose of study drug
  DOR is defined as the time between date of first response and the first occurrence of progression or death from any cause, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (24):
- United States (5):
  - University of Arizona Cancer Center - North Campus /ID# 219102, Tucson, Arizona
  - City of Hope /ID# 209786, Duarte, California
  - Hackensack Univ Med Ctr /ID# 221035, Hackensack, New Jersey
  - Lifespan Cancer Institute at Rhode Island Hospital /ID# 215418, Providence, Rhode Island
  - Prisma Health Cancer Institute-Faris Road /ID# 219076, Greenville, South Carolina
- Australia (5):
  - Royal Adelaide Hospital /ID# 223354, Adelaide, South Australia
  - St Vincent's Hospital Melbourne /ID# 222066, Fitzroy, Victoria
  - Alfred Health /ID# 214665, Melbourne, Victoria
  - Perth Blood Institute Ltd /ID# 226650, Nedlands, Western Australia
  - Royal Perth Hospital /ID# 225498, Perth, Western Australia
- France (2):
  - CHU de Nantes, Hotel Dieu -HME /ID# 215480, Nantes, Pays de la Loire Region
  - Hopital Henri Mondor /ID# 214588, Créteil
- Sheba Medical Center /ID# 214065, Ramat Gan, Tel Aviv, Israel
- Japan (4):
  - Nagoya City University Hospital /ID# 214696, Nagoya, Aichi-ken
  - National Cancer Center Hospital East /ID# 214697, Kashiwa-shi, Chiba
  - Kyushu University Hospital /ID# 220800, Fukuoka, Fukuoka
  - National Cancer Center Hospital /ID# 214801, Chuo-ku, Tokyo
- Spain (5):
  - CLINICA UNIVERSIDAD DE NAVARRA-Pamplona /ID# 217170, Pamplona, Navarra, Comunidad
  - Hospital Universitario Vall d'Hebron /ID# 214690, Barcelona
  - CLINICA UNIVERSIDAD DE NAVARRA-Madrid /ID# 214739, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 214672, Madrid
  - Hospital Universitario Virgen de la Victoria /ID# 214756, Málaga
- Taiwan (2):
  - National Taiwan University Hospital /ID# 209322, Taipei City, Taipei
  - China Medical University Hosp /ID# 209323, Taichung

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yuda J, Will C, Phillips DC, Abraham L, Alvey C, Avigdor A, Buck W, Besenhofer L, Boghaert E, Cheng D, Cojocari D, Doyle K, Hansen TM, Huang K, Johnson EF, Judd AS, Judge RA, Kalvass JC, Kunzer A, Lam LT, Li R, Martin RL, Mastracchio A, Mitten M, Petrich A, Wang J, Ward JE, Zhang H, Wang X, Wolff JE, Bell-McGuinn KM, Souers AJ. Selective MCL-1 inhibitor ABBV-467 is efficacious in tumor models but is associated with cardiac troponin increases in patients. Commun Med (Lond). 2023 Oct 25;3(1):154. doi: 10.1038/s43856-023-00380-z. PMID 37880389